CLINICAL TRIAL: NCT00535535
Title: Fructose-Induced Palmitate Synthesis in Overweight Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: The Rogosin Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: LHU-0616
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Elevated Triglycerides; Diabetes; Cardiovascular Disease
Keywords: Elevated triglycerides; Diabetes; Cardiovascular disease
MeSH Terms: conditions — Hypertriglyceridemia; Diabetes Mellitus; Cardiovascular Diseases | interventions — Fructose; Glucose

INTERVENTIONS:
Dietary Supplement: Fructose — Fructose, 0.5 g/kg
Dietary Supplement: Fructose and Glucose — Fructose:Glucose 1:1, 1 g/kg
Dietary Supplement: Fructose and Glucose — Fructose:Glucose 1:1, 2g/kg

SUMMARY:
Dietary fructose potently exacerbates the dyslipidemia associated with obesity, insulin resistance and accelerated atherosclerosis. In a randomized crossover outpatient study of 15 overweight adults, we will measure the increase over 4 hours in serum VLDL triglyceride palmitate made by the liver from each single oral dose of fructose (0.5 g/kg), fructose:glucose 1:1 (1 g/kg) or fructose:glucose 1:1 (2 g/kg). Our hypotheses are that the synthesis of palmitate from dietary fructose will be 1) greater when consumed with glucose and 2) show a dose-response. The lipogenic responses will be compared and correlated with markers of carbohydrate and lipid flux measured after fasting and post-fructose. The results will serve as a guide to the development of a new outpatient probe of the de novo lipogenic pathway in subjects who vary in their lipogenic response to oral fructose. These studies should ultimately yield valuable new information about the mechanisms linking dietary carbohydrate to elevated triglycerides, diabetes and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-75 years of age
* Body mass index (BMI) 25-35 and within 10% of maximum weight
* Willing and able to stop fish oil, psyllium, other non-prescribed vitamins/supplements for 1 week prior to study until completion of study
* Willing to not drink alcohol for 24 h before each day of blood sampling

Exclusion Criteria:

* Diabetes or other endocrine disorder, hepatitis or other liver disorder, HIV, or autoimmune disease
* Medication(s) known to affect lipids, including hormonal contraceptives
* Recent acute illness
* Gastrointestinal disease resulting in significant GI dysfunction or malabsorption
* History of fasting TG >800 mg/dl
* History of ethanol abuse (current intake >2 drinks/d) or illicit drugs
* History of severe psychiatric illness
* If female, pregnant or breastfeeding
* Participation in an investigational drug study within one month of screening
* Unusual diet or extreme level of physical activity
* Have any other condition, which in the opinion of the investigator, should prohibit the participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
A comparison of the iAUC in VLDL TG palmitate 4 hours after F:G1:1, 1g/kg, vs. 1) fructose 0.5g/kg, and 2) F:G:1:1, 2g/kg.

SECONDARY OUTCOMES:
Linear regression analysis of the relationship between the iAUC in VLDL TG palmitate after oral fructose and markers of carbohydrate and lipid flux

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C Hudgins, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

REFERENCES:
- [Derived] Hudgins LC, Parker TS, Levine DM, Hellerstein MK. A dual sugar challenge test for lipogenic sensitivity to dietary fructose. J Clin Endocrinol Metab. 2011 Mar;96(3):861-8. doi: 10.1210/jc.2010-2007. Epub 2011 Jan 20. PMID 21252253